CLINICAL TRIAL: NCT07207213
Title: Italian Adaptation and Validation of the In-person UCLA-PEERS® Model for Adolescents With Autistic Spectrum Disorder
Brief Title: SOCIAL: Adaptation and Validation of the In-person PEERS® Program for Adolescents With Autism.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS Fondazione Stella Maris (Other)
Responsible Party: Principal Investigator, Antonio Narzisi, Principal Investigator, IRCCS Fondazione Stella Maris
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Supportive Care
Other Study IDs: PEERS_ITA
Record Dates: First submitted 2024-10-09; First posted 2025-10-03 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-10

CONDITIONS: Autism Spectrum Disorder
Keywords: Autism; Adolescents; UCLA-PEERS; Social Skills; Intervention
MeSH Terms: conditions — Autism Spectrum Disorder; Autistic Disorder; Social Skills | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PEERS (Experimental): Twenty subjects will be carry out PEERS intervention
  Interventions: Behavioral: PEERS
- CONTROLS (Active Comparator): Twenty subjects will be carry out Treatment As Usual
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: PEERS — The Program for the Education and Enrichment of Relational Skills (PEERS®) is world-renowned for providing evidence-based social skills treatment to adolescents with autism spectrum disorder (ASD), attention-deficit/hyperactivity disorder (ADHD), anxiety, depression, and other socio-emotional problems.
  Other Names: TAU (TREATMENT AS USUAL)
  Arms: PEERS
Behavioral: Control — This group will also consist of children diagnosed with high-functioning ASD. However, these children will not receive PEERS therapy. Instead, they will continue their usual treatments in their local settings without participating in the PEERS therapy sessions. This group's outcomes will be compared with the experimental group to assess the effectiveness of PEERS therapy.
  Arms: CONTROLS

SUMMARY:
Autism Spectrum Disorder (ASD) falls under the category of high complexity disorders which, in most cases, accompany individuals throughout their entire life with significant impacts and costs for individuals, their families, and society at large. Adolescence is a time of increasing challenge for teenagers with ASD and their families, as it is a time to lay the foundations for the transition to adulthood but at the same time, it is a period of clear mismatch between the abilities and interests of teenagers with ASD and the expectations of their peers. It becomes increasingly difficult to initiate and maintain friendships that require social skills, communicate through social media, or make appropriate use of humor. It is in peer relationships that recognizing and applying implicit social norms is more difficult, and social errors can lead to a bad reputation, exclusion, and being bullied.

This creates the need for concrete responses through evidence-based treatment programs adapted to the Italian context. In this scenario, the Program for the Education and Enrichment of Relational Skills (PEERS®) fits in, a psychosocial intervention that falls under the category of Social Skill Training (SST) conducted in a group context, evidence-based, originating from the United States for adolescents with ASD that involves structured teaching of knowledge and skills related to social relationships.

SOCIAL has three main objectives: clinical, scientific, and social. The clinical objective is articulated in the study of the effectiveness of the in-person PEERS® program on an Italian population of adolescents with ASD (aged between 10 and 14) to respond to the evident need for a psychosocial intervention adapted to the Italian context. The scientific objective aims to identify an electroencephalographic biomarker that acts as a predictor of the efficacy of PEERS® and is specific to a particular individual profile. Finally, the social objective intends to extend the support network of adolescents with ASD through meetings with schools to train Teachers, thus parallelizing the treatment for generalization of the skills acquired during clinical treatment and also to the school context where peers play a key role.

SOCIAL aims to respond to a gap that exists in Italy for a critical age group involving teenagers with ASD, proposing an evidence-based treatment that extends to family and school contexts.

DETAILED DESCRIPTION:
Objectives SOCIAL has 3 objectives, clinical, scientific, and social in nature. At the clinical level, its objective is to test the validity and effectiveness of the in-person PEERS® program adapted to an Italian population. The main rationale is to respond to the need for a Social Skill Training adapted to the Italian context, highly acceptable, and evidence-based.

SOCIAL involves a sample of 36 adolescents with a diagnosis of autism spectrum disorder (ASD) and their parents. The subjects will be randomized into two groups (experimental group and control group). All subjects will undergo a battery of questionnaires prescribed by the PEERS® protocol administered before treatment (T0), at the end (T1), and at the 9-month follow-up from the beginning of treatment (T2). The subjects will also undergo a high-density electroencephalographic evaluation during the viewing of social content stimuli at T0, T1, and T2. The experimental group will participate in the PEERS® protocol, while the control group will undergo the usual treatment provided by the territorial reality. Test scores will be compared within-group over time (T0-T1-T2) and between groups (experimental group vs. control group).

The second scientific objective will use the electroencephalographic signal (mu rhythm desynchronization in sensorimotor regions) as a predictor of the effectiveness of PEERS®. This measure, not strictly associated with severity, becomes an implicit predictor not mediated by cognitive factors that suggest the potential effectiveness of specific treatment for a certain individual profile. As secondary outcomes, scores related to questionnaires investigating the adolescents behavior and adaptive level will also be considered.

The last social objective aims to extend the support network of adolescents with ASD to the school context through meetings that parallel the treatment in order to (1) provide supportive strategies to teachers in continuity with clinical treatment and (2) monitor the transfer of social skills in the classroom context for generalization of the skills acquired during clinical treatment.

The hypothesis is that social skills will improve following treatment for the experimental group and that the impact will also extend to other social conditions while maintaining appropriate behavior.

Methodology Participants Participants will be recruited from the Day Hospital of the IRCCS Stella Maris Foundation and residents within a distance of no more than 20/30 kilometers from the IRCCS site.

Inclusion criteria will be: (a) age between 10 and 14 years old; (b) clinical diagnosis of Autism Spectrum Disorder according to ICD-10 (WHO, 1992); (c) absence of intellectual disability (IQ over 85); (d) absence of major concomitant psychiatric disorders (e.g., schizophrenia, bipolar disorder); (e) absence of oppositional/aggressive behavior (outside of the family context); (f) difficulty in developing and/or maintaining peer relationships; (g) self-motivation to participate in treatment for both the adolescent and the family; (h) availability of a caregiver to attend regular sessions with parents and to support the participant during the program; (i) consent of parents and adolescents to participate in all evaluations and to be recorded during treatment sessions.

In accordance with the PEERS® guidelines for adolescents, the parents of candidates will undergo an initial screening through a face-to-face interview. If the initial criteria are satisfied, the parent and adolescent will be invited to an entrance interview with a psychologist who will assess the participants motivation, the risk of problem behaviors, and mental health status. During the interview, the parents availability and readiness to play the role of social coach will also be evaluated.

Once the above criteria are satisfied, the third phase will involve the administration of the Autism Diagnostic Observation Schedule, Second Edition for better phenotyping of the diagnosis, while cognitive and adaptive functioning will be evaluated using the WISC-IV (Wechsler, 2003) and Vineland-II scales. The tests will be administered by certified clinical personnel.

Instruments

Primary Outcome Measure

1. Test of Adolescent Social Skills Knowledge-Revised.
2. Quality of Socialization 2.Questionnaire-Revised.
3. Social Responsiveness Scale-2.
4. Social Skills Improvement System Rating Scales (SSiS)
5. Social Anxiety Scale (SAS)
6. Friendship Qualities Scale (FQS)
7. Piers-Harris SelfConcept ScaleSecond Edition (PHS-2)
8. Quality of Play Questionnaire (QPQ)
9. ADOS-BOSCC

Secondary Outcome Measures

1. Child Behavior Checklist 6-18 years (CBCL 6/18)
2. Youth Self Report 11-18 years (YSR 11-18)
3. Teacher Report Form 6-18 years (TRF 6-18)
4. Vineland Adaptive Behavior Scales, Second Edition (VABS-II)
5. Parenting Stress Index - IV (PSI-IV)

Electroencephalography (EEG). All subjects included in the study will undergo an approximately ten-minute electroencephalographic evaluation. The subjects will observe social content stimuli (intentional actions involving two people or basic emotional expressions). Signal analysis will focus on mu rhythm desynchronization, known in the literature as an indicator of cortical reactivity during the observation of social motor stimuli. The subjects brain reactivity will be: 1) compared to available databases of typically developing subjects during the observation of the same stimuli; 2) compared between subjects as an index of sample homogeneity at baseline; 3) for the experimental group only, the quantification of desynchronization will be considered as an index of prediction of the efficacy of the PEERS® treatment through linear and multiple regression analyses. It will be evaluated whether subjects who are more responsive to social stimuli have better prerequisites that lead to a more effective treatment. EEG recordings will be made at T0, T1, and T2 by researchers from the CNR Neuroscience Institute of Parma with proven experience in EEG signal recording and analysis. The EEG system ( BRAIN QUICK® EEG System) is a facility already available at the IRCCS Fondazione Stella Maris and will be made available to the SOCIAL project.

Experimental design Eligible study participants will be randomly assigned to either the experimental or control group. The randomization sequence will be generated using MATLAB scripts (R2021a) with a 1:1 allocation using random blocks of 2 or 4, stratified by age group. The procedure will be conducted by an independent researcher who will only know the participants identification number, age group, and sex. The latter variable is used to prevent there being only one female or male in a group. Group assignment will be concealed from participants, their parents, and personnel administering standardized tests until participants have completed baseline measures (T0).

Procedures The treatment will be conducted by PEERS® Certified Providers recognized by the Semel Institute at the University of California, Los Angeles (UCLA). The parent groups will be led by two PEERS® Certified psychologists who participated in the adaptation of the program.

Subjects in the experimental group (n=18) and their parents (n=18) will participate in one 90-minute PEERS® session per week for a total of 16 sessions. As a maximum of 6 participants per group is required, the sample will be further divided into three randomized groups. Group 1-PEERS® (n=6) will start the treatment, which will last 16 weeks, at the end of which (T1) the tests reported in the Table will be administered and the electroencephalographic activity will be recorded. Nine months after the start of the treatment, subjects will be recalled for follow-up. The procedure described above will also be used for Group 2-PEERS® (n=6) and Group 3-PEERS® (n=6). The control group sample (Group 1-CTRL, Group 2-CTRL, Group 3-CTRL) will follow the same approach, with the difference that no treatment will be proposed beyond the normal rehabilitative practices already followed.

PEERS Intervention The Program for the Education and Enrichment of Relational Skills (PEERS®) focuses on the skills necessary to initiate and maintain peer relationships, such as conversation skills, communication via electronic devices, conflict resolution, appropriate use of humor, entering and exiting peer groups, good sportsmanship, organizing get-togethers, managing disputes, changing reputation, and handling different types of bullying. The teaching techniques and materials are adapted to the learning styles of individuals with Autism Spectrum Disorder (ASD), which include visual thinking, good memory, and systematization.

In each of the 16 sessions, a therapist presents relevant skills through direct instruction, Socratic questioning, and role-playing. Participants practice skills in behavioral rehearsal exercises and receive feedback on their performance from the treatment team. Between sessions, weekly homework assignments are given, which involve practicing skills with parents and socializing with peers (e.g., talking on the phone with another group member or arranging a get-together with a friend).

Parents (or other adult family members, referred to as social coaches; in the program) participate in parallel sessions and learn how to facilitate their teens skill acquisition.

All sessions will be video recorded and treatment implementation quality will be monitored by the project supervisor (PEERS® Certified Provider). Participants treatment adherence will be monitored by recording attendance of both adolescents and social coaches, and completion rates of homework assignments.

Teens who receive PEERS® treatment will receive additional support through involvement of their school teachers. In fact, in parallel with the 16 PEERS sessions, teachers will be offered the opportunity to complete 16 sessions of Teachers coaching. Weekly tele-assistance sessions of 60 minutes will be conducted where the PEERS® Certified Provider who conducts treatment sessions with the adolescent will have a conversation with a reference teacher of the adolescent.

Ecological validity

At the end of the treatment, adolescents and parents will complete an evaluation questionnaire specifically designed for the study. The survey will include questions about participants satisfaction with various elements of the program, time burden, overall satisfaction, and willingness to recommend the program to other adolescents on the autism spectrum or their parents. The survey will also include two open-ended questions about the positive aspects of the program and those that could be improved or modified.

Results that the project aims to achieve

The efficacy of the PEERS® program for adolescents has already been confirmed by RCT studies as well as the feasibility of cultural adaptation conducted in various countries. However, the Italian adaptation is not yet available.

The expected results are: 1) to validate the efficacy of PEERS® in the Italian context; 2) to identify an electroencephalographic biomarker that acts as a predictor of treatment efficacy for a specific individual profile; 3) to provide teachers with supportive strategies in continuity with clinical treatment.

ELIGIBILITY:
Inclusion Criteria:

* (a) age between 10 and 14 years;
* clinical diagnosis of Autism Spectrum Disorder according to ICD-10 (WHO, 1992);
* absence of intellectual disability (IQ over 85);
* absence of a concomitant major psychiatric disorder (e.g., schizophrenia, bipolar disorder, psychiatric illness);
* absence of oppositional/aggressive behavior (outside the family context);
* difficulty developing and/or maintaining peer relationships;
* self-motivation to participate in the treatment of both the adolescent and the family;
* availability of a caregiver to regularly attend sessions with parents and to support the participant during the program;
* consent of the parents and the adolescent to participate in all evaluations and to be recorded during treatment sessions

Exclusion Criteria:

* Full IQ below 85;
* concomitant major psychiatric disorders

Ages: 10 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 36 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2027-01-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Test of Adolescent Social Skills Knowledge-Revised (TASSK-R) | T0 (before treatment) T1 (after 16 weeks from T0) T2 (9 months after T1)
  The TASSK-R is a self-report, criterion-referenced measure that assesses teens' knowledge about social skills taught throughout the program. It consists of 26 sentence stems in which adolescents are asked to choose from two possible answers. A higher score indicates more knowledge about social skills related to the treatment.
Quality of Socialization Questionnaire-Revised (QSQ-R) | T0 (before treatment) T1 (after 16 weeks from T0) T2 (9 months after T1)
  The QSQ-R assesses the frequency and quality of encounters of the adolescent with friends, as reported by adolescents (SQA-R) and parents (SQP-R). To verify the reliability of the report, adolescents and parents are asked to provide a list of names of the friends with whom the adolescent met. A 12-item questionnaire assesses the level of conflict during the most recent encounter with a peer, with answers given on a Likert scale.
Scala di reattività sociale-2 (SRS-2) | T0 (before treatment) T1 (after 16 weeks from T0) T2 (9 months after T1)
  The SRS-2 is a quantitative measure consisting of 65 items that assess the symptoms characteristic of autism spectrum disorders. The SRS-2 has been used in previous PEERS® program evaluations and has shown to be sensitive to treatment effects.
Social Skills Improvement System Rating Scales (SSiS) | T0 (before treatment) T1 (after 16 weeks from T0) T2 (9 months after T1)
  The SSiS is a 79-item measure that assesses general social skills general social skills and problem behaviour. It is a parent report on the behaviour of adolescents on a 4-point scale. There are standard scores are available for the general domains of social skills and problem behaviour. The SSiS has a high internal reliability.
Social Anxiety Scale (SAS) | T0 (before treatment) T1 (after 16 weeks from T0) T2 (9 months after T1)
  The SAS consists of 22 items and was developed to assess the social anxiety experienced by adolescents in the context of relationships with peers. The items are rated on 5-point Likert scale points.
Friendship Qualities Scale (FQS) | T0 (before treatment) T1 (after 16 weeks from T0) T2 (9 months after T1)
  The FQS is a self-reported measure for adolescents on the quality of best friendships. It consists of 23 items rated on a 5-point Likert scale.
Piers-Harris SelfConcept ScaleSecond Edition (PHS-2) | T0 (before treatment) T1 (after 16 weeks from T0) T2 (9 months after T1)
  The PHS-2 assesses self-esteem and self-concept. In the clinical field, it is used to determine the specific areas of conflict, coping, defense mechanisms defense mechanisms, and appropriate intervention techniques.
Quality of Play Questionnaire (QPQ) | T0 (before treatment) T1 (after 16 weeks from T0) T2 (9 months after T1)
  The QPQ consists of 12 items assessing the frequency of peer meetings during the previous month previous month and the level of conflict. This scale has been used as an outcome measure in previous studies previous studies that tested the effectiveness of social skills training.
ADOS-BOSCC | T0 (before treatment) T1 (after 16 weeks from T0) T2 (9 months after T1)
  The BOSCC (Brief Observation of Social Communication Change) is a play-based, observation tool used to measure subtle changes in social communication behaviors of individuals with autism spectrum disorder (ASD), particularly in response to early intervention. While the original BOSCC coding scheme was developed by modifying and expanding upon the Autism Diagnostic Observation Schedule (ADOS), it is a distinct outcome measure used to track changes in ASD symptoms over time. The BOSCC is considered a reliable and sensitive measure for detecting changes, even in minimally verbal individuals, and can be used across various studies and conteXT

SECONDARY OUTCOMES:
Child Behavior Checklist 6-18 years (CBCL 6/18) | T0 (before treatment) T1 (after 16 weeks from T0) T2 (9 months after T1)
  The CBCL 6-18 is widely used to assess developmental psychopathology through scales that assess syndromic, general, and emotional-behavioral dimensions according to certain DSM diagnostic categories.
Youth Self Report 11-18 years (YSR 11-18) | T0 (before treatment) T1 (after 16 weeks from T0) T2 (9 months after T1)
  The YSR was built with the aim of having a self-descriptive tool to obtain information direct information from adolescents, aged 11-18 years of age, about their skills and their behavioral and emotional problems.
Teacher Report Form 6-18 years (TRF 6-18) | T0 (before treatment) T1 (after 16 weeks from T0) T2 (9 months after T1)
  The TRF compiled by the teacher assesses the behavioural problems that an adolescent may manifest at school.
Vineland Adaptive Behavior Scales, Second Edition (VABS-II) | T0 (before treatment) T1 (after 16 weeks from T0) T2 (9 months after T1)
  VABS-II uses four specific domains: Communication, Everyday Life Skills, Socialisation, and Motor Skills. The scores of the sub-scales are summed up to obtain a composite adaptive behavior score
Parenting Stress Index - IV (PSI-IV) | T0 (before treatment) T1 (after 16 weeks from T0) T2 (9 months after T1)
  The PSI-IV consists of 120 items that assess three main stress source domains: characteristics of the adolescent, characteristics of the parent and stress situational/demographic life stress.
hd-EEG (Electrical Geodesics, Inc., Eugene, OR, USA) | T0 (before treatment) T1 (after 16 weeks from T0) T2 (9 months after T1)
  High density EEG (see

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Narzisi, PhD, Principal Investigator — IRCCS Stella Maris Foundation, Pisa (Calambrone), Italy
Locations (1):
- IRCCS Stella Maris, Calambrone, Pisa, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Laugeson EA, Frankel F, Gantman A, Dillon AR, Mogil C. Evidence-based social skills training for adolescents with autism spectrum disorders: the UCLA PEERS program. J Autism Dev Disord. 2012 Jun;42(6):1025-36. doi: 10.1007/s10803-011-1339-1. PMID 21858588
- [Background] Bramer GR. International statistical classification of diseases and related health problems. Tenth revision. World Health Stat Q. 1988;41(1):32-6. PMID 3376487
- [Background] Laugeson EA, Frankel F, Mogil C, Dillon AR. Parent-assisted social skills training to improve friendships in teens with autism spectrum disorders. J Autism Dev Disord. 2009 Apr;39(4):596-606. doi: 10.1007/s10803-008-0664-5. Epub 2008 Nov 18. PMID 19015968
- [Background] Lord C, Rutter M, DiLavore P, Risi S, Gotham K, & Bishop S (2012). Autism diagnostic observation schedule-2nd edition (ADOS-2). Los Angeles, CA: Western Psychological Services
- [Background] Wechsler D. Wechsler Intelligence Scale for Children. 4th ed. PsychCorp; San Antonio, TX, USA: 2003.
- [Background] Balboni, G., Belacchi, C., Bonichini, S., & Coscarelli, A. (2016). Vineland adaptive behavior scales. Survey interview form. Standardizzazione italiana (2nd ed.) [Vineland adaptive behavior scales. Survey interview form. Italian Standardization (2nd ed.)]. Giunti OS Organizzazioni Speciali.
- [Background] Laugeson, E. A. (2018). Quality of Socialization Questionnaire - Adolescent (QSQA- Revised). Supplement materials provided on the PEERS Certified Training Seminar, Los Angeles
- [Background] J. N. Constantino and C. P. Gruber (2012). Social Responsiveness Scale-Second Edition (SRS-2). Torrance, CA: Western Psychological Services.
- [Background] Gresham, F. M., & Elliott, S. N. (2008). Social skills improvement system: Rating scales. Bloomington, MN: Pearson Assessments
- [Background] La Greca AM, Lopez N. Social anxiety among adolescents: linkages with peer relations and friendships. J Abnorm Child Psychol. 1998 Apr;26(2):83-94. doi: 10.1023/a:1022684520514. PMID 9634131
- [Background] Bukowski, W. M., Hoza, B., & Boivin, M. (1994). Measuring Friendship Quality During Pre- and Early Adolescence: The Development and Psychometric Properties of the Friendship Qualities Scale. Journal of Social and Personal Relationships, 11(3), 471-484. https://doi.org/10.1177/0265407594113011
- [Background] Piers, E. V.
- [Background] Frankel F, Mintz J. Measuring the quality of play dates. 2011
- [Background] Achenbach, T. M., & Rescorla, L. A. (2001). Manual for the ASEBA School-Age Forms and Profiles. Burlington, VT: University of Vermont Research Center for Children, Youth, & Families.
- [Background] Abidin R.R. (2012). Parenting Stress Index, Fourth Edition (PSI-4). Lutz, FL: Psychological Assessment Resources
- [Background] Zheng S, Kim H, Salzman E, Ankenman K, Bent S. Improving Social Knowledge and Skills among Adolescents with Autism: Systematic Review and Meta-Analysis of UCLA PEERS(R) for Adolescents. J Autism Dev Disord. 2021 Dec;51(12):4488-4503. doi: 10.1007/s10803-021-04885-1. Epub 2021 Jan 29. PMID 33512626
- [Background] Shum KK, Cho WK, Lam LMO, Laugeson EA, Wong WS, Law LSK. Learning How to Make Friends for Chinese Adolescents with Autism Spectrum Disorder: A Randomized Controlled Trial of the Hong Kong Chinese Version of the PEERS(R) Intervention. J Autism Dev Disord. 2019 Feb;49(2):527-541. doi: 10.1007/s10803-018-3728-1. PMID 30143950
- [Background] Yoo HJ, Bahn G, Cho IH, Kim EK, Kim JH, Min JW, Lee WH, Seo JS, Jun SS, Bong G, Cho S, Shin MS, Kim BN, Kim JW, Park S, Laugeson EA. A randomized controlled trial of the Korean version of the PEERS((R)) parent-assisted social skills training program for teens with ASD. Autism Res. 2014 Feb;7(1):145-61. doi: 10.1002/aur.1354. Epub 2014 Jan 9. PMID 24408892
- [Background] Rabin SJ, Israel-Yaacov S, Laugeson EA, Mor-Snir I, Golan O. A randomized controlled trial evaluating the Hebrew adaptation of the PEERS(R) intervention: Behavioral and questionnaire-based outcomes. Autism Res. 2018 Aug;11(8):1187-1200. doi: 10.1002/aur.1974. Epub 2018 Aug 10. PMID 30095232
- [Background] Platos M, Wojaczek K, Laugeson EA. Effects of Social Skills Training for Adolescents on the Autism Spectrum: a Randomized Controlled Trial of the Polish Adaptation of the PEERS(R) Intervention via Hybrid and In-Person Delivery. J Autism Dev Disord. 2023 Nov;53(11):4132-4146. doi: 10.1007/s10803-022-05714-9. Epub 2022 Aug 24. PMID 36001196
- [Background] Idris S, van Pelt BJ, Jagersma G, Duvekot J, Maras A, van der Ende J, van Haren N, Greaves-Lord K. A randomized controlled trial to examine the effectiveness of the Dutch version of the Program for the Education and Enrichment of Relational Skills (PEERS(R)). BMC Psychiatry. 2022 Apr 22;22(1):293. doi: 10.1186/s12888-022-03913-3. PMID 35459118
- [Background] Rizzolatti G, Fabbri-Destro M, Cattaneo L. Mirror neurons and their clinical relevance. Nat Clin Pract Neurol. 2009 Jan;5(1):24-34. doi: 10.1038/ncpneuro0990. PMID 19129788
- [Background] Fabbri-Destro M, Avanzini P, De Stefani E, Innocenti A, Campi C, Gentilucci M. Interaction Between Words and Symbolic Gestures as Revealed By N400. Brain Topogr. 2015 Jul;28(4):591-605. doi: 10.1007/s10548-014-0392-4. Epub 2014 Aug 15. PMID 25124860